CLINICAL TRIAL: NCT04890977
Title: Engaging Pacific Islanders in Mental Health Treatment Services
Brief Title: Engaging Pacific Islanders in Mental Health Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH122641 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Talking Story (Experimental): Talking Story is a modular behavioral intervention intended to increase mental health treatment-seeking among Pacific Islanders through the use of narrative films and other culturally syntonic approaches.
  Interventions: Behavioral: Talking Story
- Wait-list control (Placebo Comparator): The wait-list control will be administered as a control arm to the active Talking Story arm.
  Interventions: Behavioral: Talking Story

INTERVENTIONS:
Behavioral: Talking Story — A culturally grounded modular intervention to increase mental health treatment-seeking among Pacific Islanders.

SUMMARY:
This study will create and pilot test a culturally grounded intervention (Talking Story) to increase mental health treatment seeking among Pacific Islanders with mental disorders (e.g., major depressive disorder, generalized anxiety disorder).

DETAILED DESCRIPTION:
For the clinical trial arm of this pilot/feasibility study, the investigators will conduct a pilottest of the culturally grounded Talking Story mental health treatment-seeking intervention with 48 Pacific Islander participants (24 intervention arm, 24 wait-list control) in preparation for larger R01 randomized wait-list controlled testing.

ELIGIBILITY:
Inclusion Criteria:

1. Of Pacific Islander or part Pacific Islander heritage,
2. Must be over 18 years of age,
3. Live in Los Angeles County or surrounding areas,
4. Fluent (oral and reading) in English,
5. Not have dual comorbidities in major depressive disorder, generalized anxiety disorder, and/or alcohol use disorder (they may have one of these disorders and still participate but not two or three).

Exclusion Criteria:

1. Do not meet inclusion criteria,
2. Are unwilling to participate,
3. Fail to provide or retracts consent,
4. Reside outside the target communities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
KAP Model | Up to 12 months
  Knowledge, Attitudes, and Practices related to seeking mental health treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UC Riverside, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided